CLINICAL TRIAL: NCT02152566
Title: Study of the Effects of Nasal High Flow Therapy as a Treatment Option for Patients With Respiratory Insufficiencies During Sleep.
Brief Title: Nasal High Flow Therapy for the Treatment of Respiratory Insufficiencies During Sleep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CIA-117
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Disordered Breathing; Congestive Heart Failure
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic PSG/PG, PSG w. nasal high flow therapy (Experimental): All patients recruited will undergo a diagnostic sleep study, either a full in laboratory attended polysomnography (PSG), or an in-home polygraphy (PG). If respiratory insufficiencies with Cheyne-Stokes respiration (CSR) are detected, these patients will undergo an overnight in laboratory attended PSG on a nasal high flow therapy device to test the primary endpoint of this study. Patients without respiratory insufficiencies after the first PSG/PG will take no further part in the trial.
  Interventions: Device: Nasal High flow therapy device

INTERVENTIONS:
Device: Nasal High flow therapy device — Nasal high flow therapy via nasal cannula.

SUMMARY:
Respiratory insufficiencies during sleep can lead to reductions in the level of oxygen in the blood during the night, which has been shown to contribute to a range of morbidities.

The purpose of this study is to assess the possibility that a nasal high flow therapy device may be able to treat respiratory insufficiencies, by stabilizing breathing and preventing reduction in blood oxygen.

Heart failure patients will be screened at a heart failure clinic, and will be asked to undergo an overnight sleep study to determine is they exhibit respiratory insufficiencies during sleep. This sleep study may be completed in the sleep laboratory (attended polysomnography, PSG) or in-home (in-home polygraphy, PG). If they are diagnosed with respiratory insufficiencies, they will be asked to attend further overnight studies to see if treatment with nasal high flow therapy can be used to stabilize breathing.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged ≥ 18 years
* Heart Failure from ischemic or non-ischemic dilated cardiomyopathy for ≥ 6 months
* Left ventricular systolic dysfunction (LVEF ≤45% by echocardiography performed within 3 months of the screening visit, or if not within 3 months, a justification provided by the cardiologist for why a repeat echocardiography is not required, for example, because the subject's condition has remained stable since their echocardiography). All echocardiography must be within a maximum of 1 year of the screening visit.
* New York Heart Association Class II or III after optimization of medical therapy
* Stable Clinical Status on stable optimal medical therapy for ≥ 1 month before entry

Exclusion Criteria:

* Unstable angina
* Myocardial infarction within the last 12 months
* Cardiac surgery within the previous 6 months
* Pregnancy
* Unwilling or unable to provide informed consent
* Uncontrolled arrhythmias
* Severe valvular heart disease
* Current/prior use of mechanical ventilation (including CPAP). At the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Vicars, PhD - Eng, Principal Investigator — Fisher & Paykel Healthcare
Locations (2):
- New Zealand (2):
  - Fisher & Paykel Healthcare Ltd., Auckland, East Tamaki
  - Middlemore Hospital, Auckland, Otahuhu

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic PSG/PG, PSG w. Nasal High Flow Therapy: All patients recruited will undergo a diagnostic sleep study, either a full in laboratory attended polysomnography (PSG), or an in-home polygraphy (PG). If respiratory insufficiencies are detected, these patients will undergo an overnight in laboratory attended PSG on a nasal high flow therapy device to test the primary endpoint of this study. Patients without respiratory insufficiencies after the first PSG/PG will take no further part in the trial.
  Nasal High flow therapy device: Nasal high flow therapy via nasal cannula.
Period: Overall Study
Arm/Group | Diagnostic PSG/PG, PSG w. Nasal High Flow Therapy
Started | 6
Completed | 3
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: From the 6 participants, 2 withdrew consent before participating in the study. 1 was lost to follow up as the participant did not turn up to his appointment.
Arm/Group | Diagnostic PSG/PG, PSG w. Nasal High Flow Therapy
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy
Description: The primary endpoint of the trial is to the efficacy of using nasal high flow therapy to stabilize breathing, as measured by the breath flow signal from PSG.
Time Frame: During 1 night of Sleep on PSG
Population: Out of 6 patient enrolled, 2 withdrew before participating in the study, 1 did not turn up to his appointment. From 3 participants who took part in the study,1 had a positive diagnosis of Cheyne-Stokes Respiration (CSR). The 1 patient who underwent treatment found the device too uncomfortable therefore no outcome measure data were available.
Arm/Group | Diagnostic PSG/PG, PSG w. Nasal High Flow Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Diagnostic PSG/PG, PSG w. Nasal High Flow Therapy
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes